CLINICAL TRIAL: NCT07249632
Title: A Phase III Trial of Telitacicept in Patients With Ocular Myasthenia Gravis
Brief Title: A Study of Telitacicept in Patients With Ocular Myasthenia Gravis (OMG)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Collaborators: Huashan Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC18-C307
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis, Ocular
MeSH Terms: conditions — Myasthenia Gravis | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telitacicept (Experimental)
  Interventions: Drug: Telitacicept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telitacicept — The dosage is administered based on the subject's age and baseline body weight, according to the following schedule:
  Subjects aged ≥18 years will receive 240 mg. Adolescent subjects aged 12 to <18 years with a body weight >50 kg will receive 240 mg. Adolescent subjects aged 12 to <18 years with a body weight between 30 kg and 50 kg (inclusive) will receive 160 mg.
  The study drug is administered once weekly (QW). Duration The double-blind treatment period will last for 24 weeks, for a total of 24 administrations of the study drug.
  Arms: Telitacicept
Drug: Placebo — The placebo contains no active ingredients. To maintain the blind, the placebo matches the active drug in all physical aspects. The placebo is administered once weekly (QW). Duration The double-blind treatment period will last for 24 weeks, for a total of 24 administrations of the placebo.
  Arms: Placebo

SUMMARY:
This is a Phase III, multicenter, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of Telitacicept for the treatment of Ocular Myasthenia Gravis (OMG).Approximately 120 eligible subjects aged 12 to 80 years with a diagnosis of OMG (Myasthenia Gravis Foundation of America [MGFA] Clinical Classification Type I) will be randomized in a 1:1 ratio to receive either Telitacicept or a matching placebo. Subjects must be on a stable standard-of-care therapy and have an MG Impairment Index (PRO) ocular score of ≥6 at screening and baseline.The study consists of a screening period of up to 6 weeks and a 24-week double-blind treatment period. The investigational product will be administered once weekly (QW) via subcutaneous injection. The dose for subjects aged ≥18 years is 240 mg. For adolescent subjects (12 to <18 years), the dose is weight-based: subjects weighing 30 to 50 kg will receive 160 mg, and subjects weighing >50 kg will receive 240 mg.The primary objective is to evaluate the efficacy of Telitacicept compared to placebo in treating OMG.The primary efficacy endpoint is the change from baseline in the MGII (PRO) ocular score at Week 24. Secondary endpoints include changes from baseline in other ocular and total scores from MGII, Myasthenia Gravis-Activities of Daily Living (MG-ADL), MG Clinical Absolute Score, and the 15-item Myasthenia Gravis Quality of Life Revised scale (MG-QOL15r). Safety and tolerability will be monitored throughout the study.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to assess the efficacy and safety of Telitacicept in subjects with Ocular Myasthenia Gravis (OMG). The study will be conducted at multiple centers.

The study duration for each subject will include a screening period of up to 6 weeks, followed by a 24-week double-blind treatment period.

Eligible subjects will be randomized in a 1:1 ratio to one of two treatment arms:

Arm 1: Telitacicept Arm 2: Placebo Randomization will be stratified by two factors: Acetylcholine Receptor (AChR) antibody status (positive vs. negative) and age (<18 years vs. ≥18 years).

Primary Objective:

To evaluate the efficacy of Telitacicept compared to placebo in the treatment of subjects with Ocular Myasthenia Gravis.

Primary Endpoint:

Change from baseline in the Myasthenia Gravis Impairment Index (Patient-Reported Outcomes) [MGII (PRO)] ocular score at Week 24.

Study Population:

A total of approximately 120 subjects will be enrolled.

Intervention:

Subjects will receive either Telitacicept or a matching placebo, administered as a once-weekly (QW) subcutaneous injection for 24 weeks. The dose will be determined based on the subject's age and body weight at baseline:

Subjects aged 12 to <18 years, with body weight 30 kg to 50 kg: 160 mg QW. Subjects aged 12 to <18 years, with body weight >50 kg: 240 mg QW. Subjects aged ≥18 years: 240 mg QW. The placebo will be identical in appearance to Telitacicept to maintain the blind.

Safety Assessments:

Safety and tolerability will be assessed through the monitoring and recording of adverse events (AEs), serious adverse events (SAEs), vital signs, physical examinations, and regular laboratory tests (hematology, serum chemistry, urinalysis). An independent Data Monitoring Committee (DMC) will be established to monitor the safety of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form.
2. Age 12 to 80 years, inclusive, male or female.
3. Body weight ≥30 kg.
4. Diagnosis of Myasthenia Gravis (MG) with documented clinical features consistent with the disease.
5. Myasthenia Gravis Foundation of America (MGFA) Clinical Classification of Type I.
6. On a stable standard-of-care (SOC) treatment regimen.

Exclusion Criteria:

1. Concomitant autoimmune diseases requiring systemic corticosteroid therapy.
2. Clinically significant laboratory abnormalities.
3. Use of other immunosuppressants (not part of the stable SOC) within 1 month prior to randomization.
4. Presence of an acute or chronic infection requiring treatment.
5. Current active hepatitis or history of severe liver disease.
6. Positive for HIV antibodies.
7. Positive for syphilis antibodies (non-specific or specific).
8. Poorly controlled diabetes mellitus, defined as HbA1c >9.0% or fasting blood glucose ≥11.1 mmol/L.
9. Subjects with thymoma (classified as ≤ Stage II for benign and ≥ Stage III for malignant according to the Masaoka staging system) .
10. Presence of uncontrolled chronic degenerative diseases, psychiatric disorders, or neurological diseases other than MG that could interfere with study assessments.
11. Other diseases causing ptosis, peripheral muscle weakness, or diplopia (e.g., Graves' ophthalmopathy, blepharospasm, progressive external ophthalmoplegia, muscular dystrophy, brainstem or cranial nerve lesions, etc.).
12. Known allergy to human-derived biological products.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the MGII (PRO) ocular score | From enrollment to the end of treatment at 24 weeks
  at Week 24

SECONDARY OUTCOMES:
Change from baseline in the MGII (PRO + PE) ocular score | From enrollment to the end of treatment at 24 weeks
  at Week 24
Change from baseline in the MG-ADL ocular score | From enrollment to the end of treatment at 24 weeks
  at Week 24
Change from baseline in the MG Clinical Absolute Score ocular score | From enrollment to the end of treatment at 24 weeks
  at Week 24
Change from baseline in the total MGII score | From enrollment to the end of treatment at 24 weeks
  at Week 24
Change from baseline in the total MG-ADL score | From enrollment to the end of treatment at 24 weeks
  at Week 24
Change from baseline in the MG-QOL15r total score | From enrollment to the end of treatment at 24 weeks
  at Week 24
Incidence and severity of adverse events | From signing of informed consent until 4 weeks after the last dose.
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

OTHER OUTCOMES:
Number and proportion of subjects who achieve MSE, defined as an MG-ADL total score of 0 or 1 | From enrollment to the end of treatment at 24 weeks
  at Week 24
Number and proportion of subjects in each MGFA-PIS category | From enrollment to the end of treatment at 24 weeks
  at Week 24
Number and proportion of subjects in each PGI-S and PGI-C category | From enrollment to the end of treatment at 24 weeks
  at Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided